CLINICAL TRIAL: NCT04183452
Title: A Comparison of Intramuscular and Subcutaneous Administration of 17-hydroxyprogesterone Caproate (17-OHPC) in Pregnancy
Brief Title: 17-OHPC in Pregnancy: IM vs SC Routes
Status: Terminated | Type: Observational
Why Stopped: Sponsor stopped study as the study drugs were withdrawn from the market
Sponsor: Steve N. Caritis, MD (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Steve N. Caritis, MD, Professor Obstetrics, Gynecology and Reproductive Science, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY19110111
Record Dates: First submitted 2019-11-19; First posted 2019-12-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Preterm Birth
Keywords: 17-hydroxyprogesterone caproate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood, 7 mL (1.5 teaspoons) will be collected from a venous catheter daily for 7 days during the pharmacokinetic (PK) study. A single sample will be collected at 3 additional times during the study: after the first injection, after 4-6 injections, and after 14-16 injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 17-Hydroxyprogesterone Caproate 250 mg IM Group: This will be an open label study and participants will not be randomized to a treatment group. The women will be prescribed 17-OHPC by their physicians because of their obstetric history. The investigators will approach pregnant women who are going to be treated with 17-OHPC and ask them to participate. The participants will select the route of administration they prefer, IM or SC. 36 participants will receive the weekly 250 mg IM dose from 16-20 weeks of pregnancy until 36 weeks or delivery.
  Interventions: Drug: 17-Hydroxyprogesterone Caproate 250 mg IM Dose
- 17-Hydroxyprogesterone Caproate 275 mg SC Group: This will be an open label study and participants will not be randomized to a treatment group. The women will be prescribed 17-OHPC by their physicians because of their obstetric history. The investigators will approach pregnant women who are going to be treated with 17-OHPC and ask them to participate. The participants will select the route of administration they prefer, IM or SC. 36 participants will receive the weekly 275 mg IM dose from 16-20 weeks of pregnancy until 36 weeks or delivery.
  Interventions: Drug: 17-Hydroxyprogesterone Caproate 275 mg SC Dose

INTERVENTIONS:
Drug: 17-Hydroxyprogesterone Caproate 250 mg IM Dose — 17-Hydroxyprogesterone Caproate is a progestin indicated to reduce the risk of preterm birth in women with a singleton pregnancy who have a history of singleton spontaneous preterm birth.
  Other Names: 17-OHPC
  Groups: 17-Hydroxyprogesterone Caproate 250 mg IM Group
Drug: 17-Hydroxyprogesterone Caproate 275 mg SC Dose — 17-Hydroxyprogesterone Caproate is a progestin indicated to reduce the risk of preterm birth in women with a singleton pregnancy who have a history of singleton spontaneous preterm birth
  Other Names: 17-OHPC
  Groups: 17-Hydroxyprogesterone Caproate 275 mg SC Group

SUMMARY:
This study will compare the plasma concentration x time curve or Area Under the Curve (AUC) and the side effects reported with 250 mg intramuscular (IM) and 275 mg subcutaneous (SC) injections of 17-hydroxyprogesterone caproate (17-OHPC).

DETAILED DESCRIPTION:
17-hydroxyprogesterone caproate (17-OHPC) is used in women with a prior preterm birth (PTB) as it reduces recurrences by a third. The drug is administered intramuscularly (IM) but that creates discomfort and in many instances requires repeated office visits as the drug is administered weekly from 16-20 weeks until 36 weeks or delivery. AMAG Pharmaceuticals obtained FDA approval to administer the drug subcutaneously (SC) based on demonstration of bioequivalence of a dose of 275 mg SC to a dose of 250 mg IM. That bioequivalence study was performed in postmenopausal women who received a single dose. This study will be performed in pregnant women with repeated injections both to demonstrate that equivalent exposure is seen and to assess the side effects and acceptance of each route of administration.

A pharmacokinetic (PK) study will be performed after participants have reached steady state (after 9 injections). Participants will receive their injections from research personnel up until the time of completion of the PK study. Home injections will be an option for all participants after the PK study is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female with documented prior birth between 16 0/7- 36 6/7 week gestation from spontaneous preterm labor or preterm premature rupture of membranes
2. Gestational age (GA) < 22 weeks, based on study determined GA (as treatment must start between 16 0/7 and 21 6/7 weeks)
3. Singleton gestation
4. Age between 18 - 45 years
5. Able to give informed consent and undergo all study procedures including a single seven day pharmacokinetic study which requires daily venipunctures and willingness to answer questions about side effects and discomfort at each study visit.

Exclusion Criteria:

1. Known major fetal anomaly or chromosomal anomalies that might affect gestational age at delivery
2. Malformation of uterus (uterine didelphus, septate uterus or bicornuate uterus)
3. Medical or obstetrical complication that might affect gestational age at delivery, such as active ulcerative colitis, liver tumors, liver disease/failure, renal disease/failure, undiagnosed vaginal bleeding unrelated to pregnancy, or hypertension requiring 2 or more agents
4. Current or history of thrombosis or thromboembolic disorders
5. Known or suspected breast cancer, other hormone-sensitive cancer, or a history of these conditions
6. Moderately severe depression (Patient Health Questionnaire-9 (PHQ-9) score ≥15, Edinburgh Postnatal Depression Scale (EPDS) score of >13, or suicidal ideation)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — study includes pregnant women
Study Population: This will be an open label study and participants will not be randomized to a treatment group. The rational for this approach is based on the expectation that the primary outcomes (AUC and side effects) will not be affected by provider or patient knowledge of or choice of treatment.
  We will approach pregnant women who are going to be treated with 17-OHPC as part of their standard of care and ask them to participate. Participants will select the route of administration they prefer, intramuscular or subcutaneous.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Compare the plasma concentration x time curve or the Area Under the Curve (AUC) of the 275 mg subcutaneous dose of 17-OHPC to the 250 mg intramuscular dose of 17-OHPC | 9 weeks after initiation (26-30 weeks gestation)
  Evaluate the difference between the plasma concentration x time curve or the Area Under the Curve (AUC) at steady state between the 250 mg dose of 17-OHPC administered intramuscularly and the 275 mg dose of 17-OHPC administered subcutaneously with an autoinjector.
Compare the severity of injection related side effects of the intramuscular and subcutaneous routes of administration of 17-OHPC | from study initiation until 36 weeks of pregnancy or delivery
  Participants will complete a Visual Analog Scale (VAS) with each injection that grades the severity of injection related side effects as none, mild, moderate or severe. This data will be used to compare the side effects of the intramuscular injections to the subcutaneous injections.
Compare the level of injection related discomfort of the intramuscular and subcutaneous routes of administration of 17-OHPC | from study initiation until 36 weeks of pregnancy or delivery
  Participants will complete a Visual Analog Scale (VAS) with each injection that grades the level of discomfort associated with the injection as none, mild, moderate or severe. This data will be used to compare the level of discomfort of the intramuscular injections to the subcutaneous injections.

CONTACTS AND LOCATIONS:
Overall Officials: Steve N Caritis, MD, Principal Investigator — University of Pittsburgh-Magee Womens Hospital
Locations (4):
- United States (4):
  - Christiana Care, Newark, Delaware
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburgh-Magee Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigator shall furnish AMAG Pharmaceuticals with the data resulting from the study, excluding any patient identifiable information. The investigator will also notify AMAG Pharmacovigilance of all serious and unexpected adverse events and provide copies of communications to and from a regulatory authority. The investigator will also provide a copy of the written consent and Institutional Review Board (IRB) approvals or renewals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified study data will be provided to AMAG within 6 months after study completion. Serious and unexpected adverse events will be reported to AMAG within three calendar days of the occurrence.